CLINICAL TRIAL: NCT07306845
Title: Veno-arterial CO2 Pressure Difference to Arterio-venous O2 Difference Ratio & Blood Lactate Levels Are Predictors of Postoperative Outcome in Whipple Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Alaa Anwar Aly Ahmed, LECTURER OF ANESTHESIA AND SURGICAL INTENSIVE CARE, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRPNO00012098
Record Dates: First submitted 2025-11-16; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Outcome; Whipple Procedures
Keywords: CO2 Pressure Difference; O2 Difference; Blood Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Predictors of Postoperative outcome in Whipple Procedures (Other): Patients undergoing Whipple surgery monitored for CO₂-derived perfusion markers (Pv-aCO₂/Ca-vO₂ ratio) & Lactate as a traditional perfusion markers.
  Interventions: Other: predictors of postoperative outcome in Whipple Procedures

INTERVENTIONS:
Other: predictors of postoperative outcome in Whipple Procedures — CO₂-Derived Parameters & Lactate as Predictors of Postoperative outcome in Whipple Procedures and the occurrence of complications

SUMMARY:
Whipple surgery is a complex abdominal procedure associated with a high risk of hemodynamic instability and splanchnic hypoperfusion leading to anastomotic leaks, delayed gastric emptying, and organ dysfunction Traditional markers (e.g., MAP, mixed venous oxygen saturation [SvO₂], lactate) are indirect, invasive and often delayed.

CO₂-derived variables (e.g., venous-to-arterial CO₂ gap [ΔCO₂], tissue CO₂ [PtCO₂], end-tidal CO₂ [EtCO₂] changes) provide earlier and more sensitive signs of microcirculatory dysfunction.

DETAILED DESCRIPTION:
Whipple surgery is a complex abdominal procedure associated with a high risk of hemodynamic instability and splanchnic hypoperfusion leading to anastomotic leaks, delayed gastric emptying, and organ dysfunction Traditional markers (e.g., MAP, mixed venous oxygen saturation [SvO₂], lactate) are indirect, invasive and often delayed.

CO₂-derived variables (e.g., venous-to-arterial CO₂ gap [ΔCO₂], tissue CO₂ [PtCO₂], end-tidal CO₂ [EtCO₂] changes) provide earlier and more sensitive signs of microcirculatory dysfunction.

The present study investigate the hypothesis that simultaneous measurement of Venous-to-Arterial CO₂ Gap Indexed to Oxygen Content Difference (Pv-aCO₂/Ca-vO₂ Ratio & blood lactate may provide one or more early markers for post-operative adverse outcome in Whipple procedure

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) undergoing open Whipple procedure under general anesthesia
* Invasive monitoring (arterial line and central venous catheter)
* Informed written consent

Exclusion Criteria:

* Emergency surgery.
* Preoperative septic shock or hemodynamic instability.
* severe pre-existing **cardiopulmonary disease (e.g., severe COPD, heart failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Venous-to-Arterial CO₂ Gap (Pv-aCO₂ = PvCO₂ - PaCO₂) | T0 baseline (After induction of anesthesia) T1 intraoperative (After major vessel dissection) T2 intraoperative (Immediately post-pancreatic resection) T3 intraoperative (After GIT anastomosis) T4 End of surgery T5 postoperative (2 hours)
  Measured via arterial and central venous blood gases sampling throughout the Whipple procedure
Arterial-Venous oxygen content difference (Ca-vO₂ = CaO₂ - CvO₂) | T0 baseline (After induction of anesthesia) T1 intraoperative (After major vessel dissection) T2 intraoperative (Immediately post-pancreatic resection) T3 intraoperative (After GIT anastomosis) T4 End of surgery T5 postoperative (2 hours) in ICU
  Measured via arterial and central venous blood gases
Veno-arterial CO2 Pressure Difference to Arterio-venous O2 Difference Ratio (Pv-aCO₂/Ca-vO₂ ratio ) | T0 baseline (After induction of anesthesia) T1 intraoperative (After major vessel dissection) T2 intraoperative (Immediately post-pancreatic resection) T3 intraoperative (After GIT anastomosis) T4 End of surgery T5 postoperative (2 hours) in ICU
  calculated by dividing the previous 2 measurements (Pv-aCO₂/Ca-vO₂ )

SECONDARY OUTCOMES:
Traditional Perfusion Markers :Lactate | T0 baseline (After induction of anesthesia) T1 intraoperative (After major vessel dissection) T2 intraoperative (Immediately post-pancreatic resection) T3 intraoperative (After GIT anastomosis) T4 End of surgery T5 postoperative (2 hours) in ICU
  Measured via arterial blood gases sampling
occurrence of Postoperative complications | within 3 days in ICU for complications, 30 days postoperatively for mortality
  • Anastomotic leak rate (pancreaticojejunostomy, hepaticojejunostomy), Delayed gastric emptying (DGE), Postoperative pancreatic fistula (POPF),
ICU length of stay | postoperative 3 days
  total ICU stay ( days)
Occurrence of post-operative complications | postoperatively within 1 month
  30-day mortality
occurrence of Organ dysfunction (AKI) | postoperatively within 3 days in ICU
  Organ dysfunction (AKI), a patient is considered to have AKI postoperatively if any one of the following occurs:
  Increase in serum creatinine ≥ 0.3 mg/dL (≥ 26.5 µmol/L) within 48 hours, OR Increase in serum creatinine to ≥ 1.5 times baseline, OR Urine output < 0.5 mL/kg/hr for ≥ 6 hours.
occurrence of postoperative complication as acute liver dysfunction | postoperatively within 3 days
  Postoperative liver dysfunction is defined as new impairment in liver function occurring after surgery, typically within the first 48-72 hours, manifested by one or more of the following: 1.Hyperbilirubinemia Total bilirubin > 2 mg/dL (34 µmol/L) OR a rise > 50% from baseline, 2.Elevated Liver Enzymes Increase in AST or ALT greater than 2-3 × upper limit of normal (ULN) Coagulopathy INR ≥ 1.5

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Anwar Abdelrahman, Dr, Principal Investigator — University of Alexandria

IPD SHARING:
Plan to Share IPD: No